CLINICAL TRIAL: NCT06272864
Title: BostonGene and Exigent Genomic INsight (BEGIN) Study: A Prospective Study of Comprehensive Molecular Testing in Advanced Cancer Patients in the Community Setting
Brief Title: BostonGene and Exigent Genomic INsight Study
Acronym: BEGIN
Status: Recruiting | Type: Observational
Sponsor: BostonGene (Industry)
Collaborators: Exigent (Unknown)
Responsible Party: Sponsor
Other Study IDs: BEGIN study
Record Dates: First submitted 2024-02-16; First posted 2024-02-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Non-small Cell Lung Cancer; Melanoma; Sarcoma
Keywords: Comprehensive Molecular Testing; BostonGene Tumor Portrait Test; Molecularly Matched Therapy; DNA and RNA Targets
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — biopsy specimen, whole blood, saliva, buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Breast cancer: Patients with locally recurrent, unresectable or metastatic breast cancer
- NSCLC: Patients with unresectable stage III or metastatic non-small cell lung cancer
- Melanoma: Patients with unresectable or metastatic melanoma
- Sarcoma: Patients with locally advanced or metastatic sarcoma

SUMMARY:
The BEGIN Study by BostonGene and Exigent Genomic INsight evaluates the efficacy of comprehensive molecular testing in advanced cancer patients. Using the BostonGene Tumor Portrait test, the study aims to identify actionable findings, assess feasibility, and determine patient enrollment in clinical trials. Four cohorts of 100 patients each will be studied over two years, focusing on treatment decisions and patient outcomes. This study seeks to demonstrate the clinical utility of genomic testing in guiding therapy for advanced cancer patients in community settings.

DETAILED DESCRIPTION:
The BEGIN Study, conducted by BostonGene and Exigent, is a prospective investigation aimed at evaluating the efficacy and feasibility of comprehensive molecular testing in advanced cancer patients within the community setting. Recent advancements in cancer treatment have led to the integration of targeted and immune-based therapies into standard practice. Recognizing the significance of genomic and molecular alterations in patient therapy selection, BostonGene has developed a high-throughput sequencing platform, the BostonGene Tumor Portrait test, which provides a comprehensive overview of tumors and their microenvironment.

The primary objectives of the study include determining the frequency of actionable findings identified by the BostonGene Tumor Portrait test, assessing the feasibility and turnaround time of comprehensive sequencing analysis, and evaluating the frequency of patient enrollment in clinical trials based on test results. Secondary objectives involve determining the frequency of patients receiving molecularly matched therapy, evaluating concordance between DNA and RNA targets, and assessing the impact of test findings on treatment decisions.

The study will involve four cohorts of patients with breast cancer, non-small cell lung cancer, melanoma, and sarcoma, each comprising 100 participants. Subjects will be identified through designated pilot sites. The study duration will be up to two years, with data collection including baseline demographics, medical history, treatment decisions, and patient outcomes.

Overall, the study aims to elucidate the clinical utility of the BostonGene Tumor Portrait test in guiding treatment decisions for advanced cancer patients in real-world community settings, with a focus on actionable findings, treatment efficacy, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed malignancy of:

Locally recurrent, unresectable, or metastatic breast cancer or; Unresectable stage III or metastatic non-small cell lung cancer or; Unresectable or metastatic melanoma or; Locally advanced or metastatic l sarcoma.

* Life expectancy > 3 months as per the treating physician
* Willingness to provide informed consent
* Living in the United States at time of enrollment
* Agree to participate in genomic and molecular profiling

Exclusion Criteria:

* not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced cancer patients
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-01-08 (Estimated); Study Completion 2028-01-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of actionable findings | 2 years
  the frequency of actionable findings identified by a comprehensive (WES/RNA) sequencing platform (BostonGene Tumor Portrait) in advanced cancer patients. Actionable findings will include: genomic findings such as fusions, single nucleotide variants (SNVs), insertion/deletion alterations (indels), copy number alterations (CNAs), tumor mutational burden (TMB), microsatellite instability (MSI), frameshifts, rearrangements, gene expression levels, genome instability and loss of heterozygosity, cell counts in TME, disease molecular type, inherited pathogenic mutations, mutational signatures, and gene isoform expression.
Test turn-around time | 2 years
  the time from consent to biopsy (or archival tissue retrieval), time from receipt of biopsy to BostonGene Tumor Portrait testing results, and total time from consent to delivery of BostonGene Tumor Portrait testing resultsTumor Portrait testing

SECONDARY OUTCOMES:
Frequency of patients who receive molecularly matched therapy | 6 months
  the frequency of patients who receive molecularly matched therapy within 6 months of undergoing genomic testing
Frequency of patients who receive molecularly matched therapy | 12 months
  the frequency of patients who receive molecularly matched therapy within 12 months of undergoing genomic testing

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Highlands Oncology Group, Rogers, Arkansas
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oncology Consultants, Houston, Texas
  - Northwest Medical Specialities, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No